CLINICAL TRIAL: NCT02715830
Title: Randomized Clinical Trial in Bellow-the-knee Angioplasty. Treatment of One or More Than One Artery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo Bruno Biagioni, Dr, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIFESP01
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Atherosclerosis of Artery
Keywords: angioplasty; infrapopliteal arteries

STUDY DESIGN:
Intervention Model Description: In this study, there is no use of other drugs, biological vaccine or combination product, but it was used two different approaches to the same problem: the renalization of the tibial arteries in patients with tissue loss. The angioplasty, that is the usual method of treatment, is done for one or more than one artery after randomization. It is phase 4 because it is an usual method of treatment (gold standard) for this disease.
Who Masked: Participant
Masking Description: The moment of randomization was after the successful accomplish of the recanalizaripn of the first artery. The used 80 sealed papers - 40 for each treatment. The nurse pick up one of the mixed papers and the procedure stops or continuous to the another artery depending on the randomization.
Oversight: Data Monitoring Committee: No

ARMS (2):
- One Artery (Experimental): In this arm after obtain the good result after the angioplasty of one artery the procedure stops
  Interventions: Procedure: Angioplasty of distal arteries
- More than one artery (Experimental): In this arm, after obtain a good result of the angioplasty of one artery, we continue trying one or two more arteries
  Interventions: Procedure: Angioplasty of distal arteries

INTERVENTIONS:
Procedure: Angioplasty of distal arteries — angioplasty of the arteries bellow-the-knee

SUMMARY:
It is a randomized study that intend to enroll 80 bellow-the-knee angioplasty procedures in which 40 procedures to treat one artery (standart) or more than one artery in the same procedure.

The aim of this study is to know if this strategy increase healing velocity and limb salvage.

ELIGIBILITY:
Inclusion Criteria:

* Occlusion of the three arteries bellow the knee previously
* Rutherford 5 - ischemic lesion of the foot
* Informative Term
* At least one patente vessel in pedal arch

Exclusion Criteria:

* allergy to aspirin, clopidogrel or contrast media
* renal impairment
* Tasc D lesion in femoral or popliteal arteries
* no undersatnting patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Time of wound healing | 1 year
  Time in days necessary to the complete healing of the wound
Limb Salvage | 1 year
  Time free of major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Marcelina Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No